CLINICAL TRIAL: NCT03759613
Title: Evaluation of Gait Symmetry in Patients With Unilateral Upper Extremity Burn Injury
Brief Title: Evaluation of Gait Symmetry in Upper Extremity Burn Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ozden Ozkal, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: GO 18/785
Record Dates: First submitted 2018-11-25; First posted 2018-11-30 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2018-11

CONDITIONS: Burn Injury
Keywords: Burn Injury; Gait Symmetry; Arm Swing
MeSH Terms: conditions — Burns | interventions — Gait Analysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Thirty subjects with unilateral upper burn injury will be included in this study. GAITRite system for gait analysis, Tampa kinesiophobia scale for kinesiophobia level, visual analog scale for pain and a scale that developed by us for arm swing will be used. Their evaluations will be made within 5 days following burn injury.
  Interventions: Other: Gait Analysis
- Control Group (Active Comparator): Thirty healthy subjects will be included in this study. GAITRite system for gait analysis, Tampa kinesiophobia scale for kinesiophobia level, visual analog scale for pain and a scale that developed by us for arm swing will be used. When their gait analysis made, they will be asked to walk their natural walking.
  Interventions: Other: Gait Analysis
- Control Grup (Restricted arm swing) (Sham Comparator): Thirty healthy subjects will be included in this study. GAITRite system for gait analysis, Tampa kinesiophobia scale for kinesiophobia level, visual analog scale for pain and a scale that developed by us for arm swing will be used. When their gait analysis made, their arms will be fixed with a bandage on their bodies. Their arm swing will be restricted.
  Interventions: Other: Gait Analysis

INTERVENTIONS:
Other: Gait Analysis — Gait Analysis: Gait analysis is not a routine assessment tool for upper extremity burn injuries. This analysis is an assessment method to estimate gait symmetry.
  Restriction arm swing: Participants in group will be restricted for arm swing using a bandage. Thus, the reciprocal arm swing will be prevented.
  Other Names: Arm Restriction

SUMMARY:
Thirty patients with unilateral burn injury, and 60 healthy subjects will be included in this study. Participants with burn injury will evaluate with the following assessment tools: Demographic data; age, gender, height, body mass index; burn characteristics; type of burn injury, degree of burn injury, localization of burn injury and total burn surface area will be recorded. Gait parameters (step length, stride length, base support, step time, cycle time, cadence, velocity, single support, double support, swing ( % of gait cycle) and stance (% of gait cycle). will be recorded via computerized system. And gait symmetry will be calculated via formule. Participants' kinesiophobia level will be evaluated with Tampa kinesiophobia scale. Their pain will be assessed by visual analog scale. Their arm swing will be evaluated by a scale.

DETAILED DESCRIPTION:
Thirty individuals with lower extremity burn injury and sixty healthy subjects will be included in this study. Participants with burn injury will be included if they are aged of 18-50, able to walk independently at least 10 meters. Healthy subjects will be included if there are no orthopedic, neurological or musculoskeletal disorders that affect gait.

1. Group: 30 Patients with burn injury
2. Group: 30 healthy subjects (When evaluating the gait analysis, their arm will not be restricted (Their natural walking)
3. Group : 30 healthy subject (When evaluating the gait analysis, their arm will be restricted )

Participants will evaluate with the following assessment tools: Demographic data; age, gender, height, body mass index; burn characteristics; type of burn injury, degree of burn injury, localization of burn injury and total burn surface area will be recorded.

All subjects' gait analysis will be conducted via GAITRite (computerized) system.

GAITRite system for gait parameters (step length, stride length, base support, step time, cycle time, cadence, velocity, single support, double support, swing ( % of gait cycle) and stance (% of gait cycle), Tampa Kinesiophobia scale for kinesiophobia level, visual analog scale for pain, a scale that developed by us for arm swing will be used.

These evaluations will be applied one time for participants. These evaluations will be made within 5 days following burn injury.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of upper extremity burn injury
* must be able to walk independently
* Control group consists of healthy adults with the similar demographic characteristics as experimental group.

Exclusion Criteria:

* Walking with assist device
* Having a visual deficits
* Having an orthopedic problems that affect gait
* Having a neurological disorders
* Having a musculoskeletal disorders that affect gait
* Having an undergone orthopedic surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Gait Speed | through study completion, an average of 5 months
  It is measured by computerized gait analysis system. Speed is the distance walked per unit of time. It is determined in centimeters per second (cm/sec)
step length | through study completion, an average of 5 months
  It is measured by computerized gait analysis system. Difference in position between the feet at heel strike, in the direction of forward motion. The unit of measure is centimeters. It is calculated both right and left foot.
Swing phase | through study completion, an average of 5 months
  It is measured by computerized gait analysis system. Swing Phase,which accounts for 40% of a single gait cycle, the phase during which the foot is not in contact with the ground. It is expressed in seconds (sec) and as a percentage of the gait cycle of the same foot. It is calculated both right and left foot.
Stance Phase | through study completion, an average of 5 months
  It is measured by computerized gait analysis system.The gait phase that lasts from heel strike to toe off, which accounts for 60% of a single gait cycle. It is expressed in seconds (sec) and as a percentage of the gait cycle of the same foot. It is calculated both right and left foot.
Single Support | through study completion, an average of 5 months
  It is measured by computerized gait analysis system. Only one foot in contact with the floor. It is expressed as a percentage of the gait cycle. It is calculated both right and left foot.
Double Support | through study completion, an average of 5 months
  It is measured by computerized gait analysis system. Boot feet in contact with the floor. It is expressed as a percentage of the gait cycle. It is calculated both right and left foot.
Gait symmetry index | through study completion, an average of 5 months
  It's calculated in order to evaluate symmetry for bilateral parameters of gait. The value of symmetry index =0 equals full symmetry. Minimum score is 0 indicates perfect symmetry. Maximum score is endless. The higher score is indicated the more asymmetrica gait pattern.
Cadence | through study completion, an average of 5 months
  It is measured by computerized gait analysis system. Rhythm expressed in steps per second.
Base support | through study completion, an average of 5 months.
  It is measured by computerized gait analysis system. It is the distance between two linescutting feet equal halves. The unit of measure is centimeters.

SECONDARY OUTCOMES:
Tampa Kinesiophobia Scale | through study completion, an average of 5 months
  This scale consists of a 17-item self-report questionnaire that measures the fear of re-injury because of movement. Items are scored on a 4-point Likert scale ranging from 1 "strongly disagree" to 4 "strongly agree". The total scores for scale range from 17 to 68. Maximum score means higher level of kinesiophobia.
Pain severity | through study completion, an average of 5 months
  Pain severity was assessed by visual analogue scale. This scale score range from "no pain=0 point " to "worst imaginable pain=10 points" for intensity. Maximum point means worst pain severity.
Arm swing | through study completion, an average of 5 months
  Arm swing will be evaluated with an arm swing scale. Arm swing scale consists of a 5 item questions for each side (left arm-right arm). Totally, scale consist of 10 questions. Scale score range from "10 points: indicates normal arm swing" to "0 points: indicates totally restricted arm swing. Maximum score means best arm swing.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozkal, PhD, PT, Principal Investigator — Hacettepe University
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)